CLINICAL TRIAL: NCT06899087
Title: DEciphering CIrculating SIgnatures Of Infected Pancreatic Necrosis
Status: Recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: DECISION
Record Dates: First submitted 2025-03-18; First posted 2025-03-27 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Acute Pancreatitis
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — venous blood samples will be collected
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: participants locally through the University of Minnesota and the M Health Fairview system before the two-week mark following acute pancreatitis onset
  Interventions: Other: not interventional

INTERVENTIONS:
Other: not interventional — This is an observational study

SUMMARY:
The purpose of the study is to identify novel blood-based biomarkers for prediction and diagnosis of infected pancreatic necrosis (IPN) in patients with necrotizing pancreatitis (NP).

Acute pancreatitis (AP) is the leading cause of gastrointestinal hospital admissions, accounting for over 300,000 emergency department visits annually and imposing a significant socio-economic burden. It is an acute inflammatory condition of the pancreas characterized by damage to the acinar cells, which triggers an inflammatory response and causes widespread systemic damage. In about 20% of cases, the disease progresses to necrotizing pancreatitis (NP), a severe form characterized by tissue necrosis. NP poses serious health risks, especially when the necrotic tissue becomes infected, leading to infected (peri-)pancreatic necrosis (IPN), which is associated with secondary organ failure (OF), sepsis, and mortality rates as high as 40%. While patients with sterile (peri-)pancreatic necrosis (SPN) can often be managed conservatively, those with IPN typically require antibiotics and therapeutic interventions such as endoscopic drainage or surgery.

Timely recognition and treatment of IPN are crucial for improving patient outcomes, yet current diagnostic methods based on clinical symptoms and routine lab markers lack the specificity to reliably distinguish SPN from IPN in the early stages. Furthermore, while multifactorial scoring systems like Ranson, Imrie, and APACHE II predict necrosis and overall severity in AP, they are not accurate for identifying IPN or predicting mortality in NP. The diagnostic gap delays appropriate treatment, allowing the infection to advance and limiting available therapeutic options. The growing incidence and significant impact of AP and NP in the general population underscore the urgent need to better understand IPN pathophysiology and to develop specific diagnostic biomarkers that can improve prognosis, guide therapeutic decisions, and enhance patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged >18 years.
* Diagnosis of NP based on CECT.

Exclusion Criteria:

* recurrent AP
* pancreatic cancer
* pregnancy, lactation
* solid organ transplant
* immunodeficiency disorders like AIDS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (>18 years) patients with a diagnosis of NP based on contrast-enhanced computed tomography (CECT) after 2 weeks from AP onset at the University of Minnesota will be included. The study does not restrict enrollment based on sex, gender, race, ethnicity, or other demographic factors. Non-demographic factors such as social determinants of health, socioeconomic status, and comorbidities will be considered in the study analysis.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Understand immune-metabolic dynamics in NP | 3 months
  by assessing pro- and anti-inflammatory cytokines, immune response of peripheral blood mononuclear cells (PBMCs), and plasma metabolites
Identify novel biomarkers | 3 months
  Using venous blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Guru Trikudanatham, MD, Principal Investigator — University of Minnesota; Petr Vanek, MD, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States